CLINICAL TRIAL: NCT01160094
Title: Clinical Outcomes on ErbB2+ MBC Patients Treated With Lapatinib-Capecitabine After Trastuzumab Progression: Role of Early Versus Late Switch to Lapatinib-Capecitabine (TYCO)
Brief Title: Role of Early Versus Late Switch to Lapatinib-Capecitabine (TYCO)
Acronym: TYCO
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 113780
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Cancer
Keywords: Trastuzumab; Metastatic Breast Cancer; Breast Cancer; Observational Study; Lapatinib
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: ErbB2+ metastatic breast cancer patients
  Interventions: Drug: Treatment

INTERVENTIONS:
Drug: Treatment — patients treated with Lapatinib-Capecitabine after Trastuzumab Progression

SUMMARY:
It will be conducted as an international multicenter prospective observational cohort study in a population of ErbB2 positive metastatic breast cancer patients, whose disease has progressed after trastuzumab-containing regimen, comparing outcomes in two groups: Group 1: patients receiving Lapatinib-capecitabine immediately after 1st Trastuzumab progression (second line treatment), and Group 2: patients receiving Lapatinib-capecitabine after 2 or more lines of treatment after 1st trastuzumab progression (third line or greater).

DETAILED DESCRIPTION:
Lapatinib in combination with capecitabine is a standard of care treatment for ErbB2+ metastatic breast cancer (MBC) patients who have progressed after anthracyclines, taxanes and trastuzumab treatment. Results from the lapatinib pivotal trial showed that the addition of lapatinib to capecitabine increased median time to progression (TTP) even among heavily pre-treated patients (median of 4 prior lines of therapy). A recent ad hoc subset analysis of this trial suggested that earlier administration of lapatinib-capecitabine in MBC patients who progress after trastuzumab may produce better clinical outcomes. The TYCO study was designed to evaluate if early switch to lapatinib-capecitabine in patients with ErbB2+ MBC who have progressed on trastuzumab-containing regimen improves TTP in comparison with a later start (after several lines of therapy). Secondary objectives include Overall Response Rate (ORR), 1 year Overall Survival (OS), and description of reported serious adverse events. This is an international, multicenter, prospective, observational (non-interventional) study in 269 ErbB2+MBC patients whose disease has progressed after treatment with trastuzumab. Two cohorts will be compared; Group 1: patients receiving lapatinib-capecitabine immediately after first trastuzumab progression, and Group 2: patients receiving lapatinib-capecitabine after two or more lines of treatment after first trastuzumab progression. Eligibility criteria include females aged 18 or more with confirmed ErbB2+ MBC who have progressed after a previous trastuzumab-containing regimen, eligible to start standard therapy with lapatinib-capecitabine at approved conventional doses, as per local label approval. The study duration is of 12 months with data collection at baseline and approximately every 3 months thereafter. Patient evaluations will be conducted per standard patient care in each center and TTP will be determined by the treating physician (clinically or radiologically). Enrollment started in February 2010 and completion of accrual is estimated for December 2011.

ELIGIBILITY:
* Women with ErbB2+ MBC (ErbB2 expression confirmed by immunohistochemistry or FISH/CISH, either in the primary tumor or in the metastasis, according to the institution's common practice);
* Older than 18 years old;
* Have received prior treatment with trastuzumab-containing regimen for ErbB2+ breast cancer;
* Progressing after trastuzumab-containing regimen either used for the treatment of metastatic disease or progressing after adjuvant /neoadjuvant trastuzumab treatment;
* Eligible to start standard treatment with Lapatinib-capecitabine at conventional doses, OR receiving standard treatment with
* Lapatinib-capecitabine at conventional doses, for no longer than 10 weeks from the start of the treatment to the date of inclusion in the study;
* Signed consent to participate and release information for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases of ErbB2 positive metastatic breast cancer, receiving approved standard treatment with lapatinib-capecitabine, after trastuzumab-containing regimen progression in community setting. Patients from private and public settings.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2010-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Time to disease progression | One year
  the time from the date of start of Lapatinib capecitabine treatment until date of documented disease progression by the treating physician

SECONDARY OUTCOMES:
Overall Response Rate | One year
  the percentage of patients showing complete response (CR) and partial response (PR) to the given treatment.
Overall survival | measured at the end of follow-up
  the time from the start of lapatinib capecitabine treatment until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Colombia (5):
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Bucaramanga
  - Novartis Investigative Site, Medellín
  - Novartis Investigative Site, Pasto
  - Novartis Investigative Site, Pereira
- Saudi Arabia (3):
  - Novartis Investigative Site, Dammam
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh